CLINICAL TRIAL: NCT00271752
Title: The Procalcitonin and Survival Study - A Multicentre Single Blinded Randomized Controlled Trial to Investigate if Treatment Guided by Daily Procalcitonin Measurements Can Reduce Mortality in the Intensive Care Unit
Brief Title: The Procalcitonin and Survival Study
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Procalcitonin Study Group (Other)
Collaborators: Copenhagen HIV Programme (Other Government); Danish Research Agency (Other); Hvidovre University Hospital (Other)
Responsible Party: Jens-Ulrik Jensen/ MD, Copenhagen HIV Programme, Faculty of Health Sciences, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PASS
Record Dates: First submitted 2006-01-01; First posted 2006-01-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Localized Infection; Sepsis; Multiple Organ Failure
Keywords: Procalcitonin; Sepsis; Intensive Care Unit; Sepsis and Complications; Organ Failure
MeSH Terms: conditions — Focal Infection; Sepsis; Multiple Organ Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCT guided (Experimental): Procalcitonin guided treatment of infections in the ICU. Intervention: Intensification of antibiotics, surgery, microbiologic testing and diagnostic imaging, when Procalcitonin levels are increasing
  Interventions: Procedure: Earlier therapeutic changes regarding infection
- Control (Sham Comparator): These patients receive "Standard of Care" which is the recommended treatment in the given ICU
  Interventions: Procedure: Earlier therapeutic changes regarding infection

INTERVENTIONS:
Procedure: Earlier therapeutic changes regarding infection — For every day Procalcitonin levels increase in the intervention group, antibiotics, surgery, diagnostic imaging and microbiologic testing is intensified

SUMMARY:
This is a randomised, single blinded, multicentre trial to evaluate whether daily procalcitonin (PCT) measurements and immediate diagnostic and therapeutic responses to abnormal values and day-to-day changes can reduce the mortality of critically ill patients in the Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
Sepsis and complications to sepsis are major causes of mortality in critically ill patients. Rapid treatment of sepsis is of crucial importance for survival of patients. In the ICU, the infectious status of the patient is often difficult to assess because symptoms cannot be expressed (unconscious or sedated patients) and signs may present atypically because of immunologic incompetence and masking by the drugs given and thermo-therapy. Biological and biochemical markers of inflammation (White Blood Cells (WBC), C-reactive protein) may often be influenced by other parameters than infection, such as: trauma, surgery, other types of inflammation such as rheumatoid diseases (C-reactive protein) and gluco-corticosteroid treatment (WBC), and may be unacceptably slowly released after progression of an infection. At the same time, lack of a relevant antimicrobial therapy in an early course of infection may be fatal for the patient.

For these reasons, in the clinical setting, it is often necessary to initiate or adjust antimicrobial therapy on an unsure ground and the relevant therapy may in some situations be delayed for important hours or even days. Specific and rapid markers of bacterial infection have been sought for use in the ICU. Mortality in critically ill patients increases gravely when Procalcitonin levels increase from day to day (own submitted, though yet unpublished data). Low PCT levels have been shown to effectively rule out sepsis.

However, no randomised controlled trials have been conducted to show if mortality in critically ill patients can be reduced by using a strategy of daily standardised Procalcitonin measurements as an early detector of serious bacterial infection. Therefore evidence is presently not sufficient to introduce daily consecutive Procalcitonin measurements to guide the diagnostic and therapeutic management of patients admitted to the ICU .

The rationale for this trial is to assess the ability of daily Procalcitonin measurements to reduce the mortality of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

Fulfilment of all of the following three criteria:

1. Male or female, aged > 18 years of age.
2. Admitted to the participating Intensive Care Units (ICUs) at the following hospitals: Hvidovre Hospital, Bispebjerg Hospital, Amager Hospital, Herlev Hospital, Glostrup Hospital, and Gentofte Hospital
3. Ability to understand and provide written informed consent to participate in this trial; or ability to understand and provide oral informed consent in the presence of at least one impartial witness who should sign and personally date the consent form; or the subject's legally acceptable representative can understand and provide written informed consent if the subject is not capable of this because of the present mental or physical condition of the subject.

Exclusion Criteria:

A subject will NOT be eligible for inclusion in this trial if any of the following criteria apply:

1. Subjects with known hyperbilirubinaemia (> 0.4 mg/ml) or hypertriglyceridaemia (> 10 g/l) since this can interfere with measurements. If subjects with unknown status on these points are included and have PCT measurements, the measuring equipment will detect these conditions.
2. Subjects suffering from a blood disorder, where daily sampling of 7 ml of blood for a maximum of 28 days (210 ml distributed on 28 days) will be an inconvenience or a potential risk, which could compromise the safety of the subject.
3. Subjects who are pregnant or breast feeding

The a priori probability of surviving with the normal recommended diagnostics and treatment with the presently available means to detect infections and, on the other hand, the normal diagnostics and treatment together with daily procalcitonin measurements and prompt clinical reaction should be equal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
mortality/survival | 28 day

SECONDARY OUTCOMES:
mortality/survival | 60 day
mortality/survival | 90 day
mortality/survival | 120 day
mortality/survival | 180 day
Consumption of antimicrobial chemotherapy | 28 day
Prevalence of complications to infection: sepsis | 28 day
severe sepsis | 28 day
septic shock | 28 day
Multi Organ Dysfunction Syndrome | 28 day
Disseminated Intravascular Coagulation | 28 day
use of diagnostic imaging during admission to the ICU | 28 day
Quality of life post-ICU | 180 day

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik S Jensen, MD, PhD, Study Director — Dept. of Clinical Microbiology, Hvidovre University Hospital & Copenhagen HIV Programme (CHIP), Faculty of Health Sciences, University of Copenhagen
Locations (9):
- Denmark (9):
  - Intensive Care Unit, Århus Sygehus, Nørrebrogade, Aarhus, Central Jutland
  - Skejby Sygehus, Skejby, Århus, Central Jutland
  - Intensive Care Unit, Bispebjerg Hospital, Copenhagen NV, Copenhagen
  - Intensive Care Unit, KAS Gentofte, Gentofte Municipality, Copenhagen
  - Intensive Care Unit, KAS Glostrup, Copenhagen University Hospital, Glostrup Municipality, Copenhagen
  - Intensive Care Unit, Herlev Hospital, Herlev, Copenhagen
  - Intensive Care Unit 542, Hvidovre Hospital, Copenhagen University Hospital, Hvidovre, Copenhagen
  - Intensive Care Unit, Hilleroed Sygehus, Hilleroed, Frederiksborg County
  - Roskilde Sygehus, Roskilde, Region Sjælland

REFERENCES:
- [Derived] Holm FS, Sivapalan P, Seersholm N, Itenov TS, Christensen PH, Jensen JS. Acute Lung Injury in Critically Ill Patients: Actin-Scavenger Gelsolin Signals Prolonged Respiratory Failure. Shock. 2019 Sep;52(3):370-377. doi: 10.1097/SHK.0000000000001279. PMID 30339635
- [Derived] Jensen JS, Itenov TS, Thormar KM, Hein L, Mohr TT, Andersen MH, Loken J, Tousi H, Lundgren B, Boesen HC, Johansen ME, Ostrowski SR, Johansson PI, Grarup J, Vestbo J, Lundgren JD; Procalcitonin And Survival Study (PASS) Group. Prediction of non-recovery from ventilator-demanding acute respiratory failure, ARDS and death using lung damage biomarkers: data from a 1200-patient critical care randomized trial. Ann Intensive Care. 2016 Dec;6(1):114. doi: 10.1186/s13613-016-0212-y. Epub 2016 Nov 21. PMID 27873291
- [Derived] Johansen ME, Johansson PI, Ostrowski SR, Bestle MH, Hein L, Jensen AL, Soe-Jensen P, Andersen MH, Steensen M, Mohr T, Thormar K, Lundgren B, Cozzi-Lepri A, Lundgren JD, Jensen JU. Profound endothelial damage predicts impending organ failure and death in sepsis. Semin Thromb Hemost. 2015 Feb;41(1):16-25. doi: 10.1055/s-0034-1398377. Epub 2015 Jan 15. PMID 25590523
- [Derived] Johansen ME, Jensen JU, Bestle MH, Hein L, Lauritsen AO, Tousi H, Larsen KM, Loken J, Mohr T, Thormar K, Johansson PI, Cozzi-Lepri A, Lundgren JD. The potential of antimicrobials to induce thrombocytopenia in critically ill patients: data from a randomized controlled trial. PLoS One. 2013 Nov 28;8(11):e81477. doi: 10.1371/journal.pone.0081477. eCollection 2013. PMID 24312305
- [Derived] Jensen JU, Hein L, Lundgren B, Bestle MH, Mohr T, Andersen MH, Thornberg KJ, Loken J, Steensen M, Fox Z, Tousi H, Soe-Jensen P, Lauritsen AO, Strange DG, Reiter N, Thormar K, Fjeldborg PC, Larsen KM, Drenck NE, Johansen ME, Nielsen LR, Ostergaard C, Kjaer J, Grarup J, Lundgren JD; Procalcitonin And Survival Study (PASS) Group. Kidney failure related to broad-spectrum antibiotics in critically ill patients: secondary end point results from a 1200 patient randomised trial. BMJ Open. 2012 Mar 11;2(2):e000635. doi: 10.1136/bmjopen-2011-000635. Print 2012. PMID 22411933
- [Derived] Jensen JU, Hein L, Lundgren B, Bestle MH, Mohr TT, Andersen MH, Thornberg KJ, Loken J, Steensen M, Fox Z, Tousi H, Soe-Jensen P, Lauritsen AO, Strange D, Petersen PL, Reiter N, Hestad S, Thormar K, Fjeldborg P, Larsen KM, Drenck NE, Ostergaard C, Kjaer J, Grarup J, Lundgren JD; Procalcitonin And Survival Study (PASS) Group. Procalcitonin-guided interventions against infections to increase early appropriate antibiotics and improve survival in the intensive care unit: a randomized trial. Crit Care Med. 2011 Sep;39(9):2048-58. doi: 10.1097/CCM.0b013e31821e8791. PMID 21572328
- [Derived] Jensen JU, Lundgren B, Hein L, Mohr T, Petersen PL, Andersen LH, Lauritsen AO, Hougaard S, Mantoni T, Bomler B, Thornberg KJ, Thormar K, Loken J, Steensen M, Carl P, Petersen JA, Tousi H, Soe-Jensen P, Bestle M, Hestad S, Andersen MH, Fjeldborg P, Larsen KM, Rossau C, Thomsen CB, Ostergaard C, Kjaer J, Grarup J, Lundgren JD. The Procalcitonin And Survival Study (PASS) - a randomised multi-center investigator-initiated trial to investigate whether daily measurements biomarker Procalcitonin and pro-active diagnostic and therapeutic responses to abnormal Procalcitonin levels, can improve survival in intensive care unit patients. Calculated sample size (target population): 1000 patients. BMC Infect Dis. 2008 Jul 13;8:91. doi: 10.1186/1471-2334-8-91. PMID 18620598